CLINICAL TRIAL: NCT01427556
Title: CCRC: The Hormonal and Behavioral Impact of Eating Breakfast
Brief Title: The Hormonal and Behavioral Impact of Eating Breakfast
Acronym: FL-74
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WHNRC 213098-1
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Eating Behavior
Keywords: Food intake; Breakfast eating
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and saliva samples will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breakfast Eaters: Women who self-report eating breakfast regularly.
- Non-Breakfast Eaters: Women who self-report skipping breakfast regularly.

SUMMARY:
This study is exploring the relationship between food intake behavior and the hypothalamic-pituitary axis (HPA) in women who regularly skip breakfast compared to women who regularly eat breakfast.

DETAILED DESCRIPTION:
Healthy women will be studies in a cross-sectional fashion to examine the metabolic, hormonal and behavioral factors associated with breakfast skipping.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women (as determined by self-report of menstrual history and confirmation with plasma FSH)
* 20 to 45 years old,
* BMI less than 40 kg/m2
* Stable body weight (fluctuation of less than ± 3%) for past 3 months.
* Breakfast eaters: defined as eating at least 15% of total daily energy intake at a meal between 0400-1000 h at least 6 days/week.
* Breakfast skippers: defined as eating no foods or beverages between 0400-1000h at least 4 days/week or only taking beverages (no solid food) containing less than ~100 kcal.

Exclusion Criteria:

* Erratic/intermittent breakfast eating
* Currently pregnant or lactating
* Shift workers/diagnosed sleep disorders
* Use of tobacco products
* Use of non-prescription drugs/hormone replacement/steroid-based medications
* Diagnosed endocrine, metabolic, or digestive disorder
* Hemoglobin <11 g/dl
* Plasma Glucose >120 mg/dl

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One hundred and twenty pre-menopausal women, aged 20 to 45y, who report eating breakfast regularly or skipping breakfast regularly.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Food Intake Behavior | week 6
  The goal is to explore the relationship between food intake behavior and the hypothalamic-pituitary axis (HPA) in a group of women who regularly skip breakfast and in another group of women who regularly eat breakfast.

SECONDARY OUTCOMES:
Markers of nutrient metabolism | week 6
  Blood glucose, insulin, lipids, and metabolic hormones will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Keim, PhD, Principal Investigator — WHNRC, ARS, University of California Davis
Locations (1):
- Western Human Nutrition Center, University of California Davis, Davis, California, United States

REFERENCES:
- [Derived] Forester SM, Widaman AM, Krishnan S, Witbracht MG, Horn WF, Laugero KD, Keim NL. A Clear Difference Emerges in Hormone Patterns Following a Standard Midday Meal in Young Women Who Regularly Eat or Skip Breakfast. J Nutr. 2018 May 1;148(5):685-692. doi: 10.1093/jn/nxy020. PMID 29897486